CLINICAL TRIAL: NCT02893176
Title: Potential Therapy With MACITENTAN in the Treatment of Chronic Lung Allograft Dysfunction (CLAD) After Lung Transplantation
Brief Title: Macitentan in the Treatment of Organ Rejection After Lung Transplantation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-001710
Record Dates: First submitted 2016-03-09; First posted 2016-09-08 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Lung Transplant Rejection
Keywords: Lung Transplant; Macitentan; CLAD; BOS; bronchiolitis obliterans; chronic lung allograft dysfunction; Organ Rejection
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 10mg will be administered one time daily
  Interventions: Drug: placebo (for macitentan)
- Active (Active Comparator): 10mg macitentan will be administered one time daily
  Interventions: Drug: macitentan

INTERVENTIONS:
Drug: macitentan
  Other Names: Opsumit
  Arms: Active
Drug: placebo (for macitentan)
  Arms: Placebo

SUMMARY:
Potential therapy with MACITENTAN in the treatment of Chronic Lung Allograft Dysfunction (CLAD) after Lung Transplantation. Pilot Study, Double-blind, "ADD-ON Therapy" with MACITENTAN to "usual standard of care immunosuppressive therapies" after lung transplantation for established BOS Stages I or II versus a "matched control group" who receive "usual standard of care immunosuppressive therapies" alone, results in a decrease in the Primary Endpoint: "rate of decline" in "Forced Expiratory Volume-1 sec (FEV1) versus time" while Secondary Endpoints including: differences in Six minute walk distance (6MWD), BORG Score, corrected single-breath diffusing capacity (DCO corrected) at time intervals of 1, 3, 6 months on therapy. Specific biomarkers for BOS, including inflammatory chemokines, which are routinely collected in the context of post-transplant "surveillance" will be analyzed. Chemokines which our group has previously described in the pathogenesis of the continuum of "acute-to-chronic lung allograft rejection", have included both C-C (CCL2, CCL5) and CXC (CXCL9, CXCL10, CXCL11) chemokines as determined in bronchial-alveolar lavage (BAL).

DETAILED DESCRIPTION:
Preliminary studies employing a "rat tracheal allograft transplant model" have demonstrated amelioration of the fibrous airway obliteration associated with blockade of the renin-angiotension and the endothelin system implementing the ERA antagonist, BOSENTAN (100 mg/kg). Clinical studies have indeed demonstrated that the mitogenic and profibrotic peptide, ET-1, may represent a potential biomarker in clinical BOS. Detection of levels of ET-1 mRNA were significantly increased in the lung allografts of those with versus those without BOS at 3 and 12 months post-transplantation while ET-1 concentrations were significantly elevated both in serum and bronchoalveolar lavage fluid (BALF) from patients with BOS. Additional studies have further demonstrated a pronounced inhibitory effect elicited by chronic ET(A) receptor blockade in the absence of immunosuppressive therapy, on both plasma levels and transcriptional regulation of inflammatory chemokines in a rat heterotopic heart transplant model of chronic rejection .

MACITENTAN, a novel, competitive ERA with significantly slower receptor dissociation kinetics than currently approved ERAs, may represent a renewed hope for patients suffering from progressive CLAD post-transplantation. The efficacy of MACITENTAN was not realized in the exploratory Phase II MUSIC Trial for IPF for the primary endpoint measure of forced vital capacity (FVC), nevertheless, mechanistic disparities in the pathobiology of CLAD versus IPF, therefore should not preclude a separate therapeutic trial. Further, in vitro treatment with MACITENTAN and its major metabolite (ACT-132577) decreases alpha smooth muscle actin elaboration by dermal fibroblasts in systemic sclerosis fibrotic skin lesions, therefore offering significant promise for potential disease modulation. Most importantly, the MUSIC Trial has further demonstrated the "clinical safety" of this pharmacologic therapy in 178 patients with IPF with mean drug exposure of approximately 14 months and without statistical differences in incidence of abnormal liver function studies. Recent pharmacokinetic studies of MACITENTAN have suggested no "clinically significant" drug-drug interaction with respect to Cytochrome P4503A4 for concurrent post-transplant immunosuppressive type therapies, such as cyclosporine, tacrolimus and mycophenolate mofetil; while insignificant interaction with the frequently implemented "azole-type antibiotics" was also observed.

ELIGIBILITY:
Inclusion Criteria:

* UCLA unilateral or bilateral lung transplant recipients, ages: 21-65 years.
* Females of child bearing age who could become pregnant, must implement appropriate contraception per FDA requirement for "ERA medical treatment" with mandatory MONTHLY monitoring of urine or serum pregnancy tests.
* No concurrent clinically significant chronic liver disease
* Screening echocardiogram (performed as usual post-transplant standard of care) with LVEF>40%, only "Grade I" or less for "LV diastolic dysfunction".
* Non-intubated, fully ambulatory patients who can perform respiratory maneuvers for office Spirometry and DCO and 6MWD (no tracheostomy).
* Total of 20 patients with BOS Stage I or II, randomized double-blind to 'standard of care + placebo" versus "standard of care + MACITENTAN" Groups.
* Laboratory "safety studies" are already routinely monitored in the context of post-transplant patients' chronic immunosuppressive regimen and include: comprehensive metabolic panel, tacrolimus trough level, B-type natriuretic peptide (BNP), CBC + platelet count.
* "Physiologic" outcomes for this study are already considered "standard of care" for lung transplant recipients that include: Office-based Spirometry pre- and post-bronchodilator, corrected DCO, six minute walk distances + BORG score assessments (6MWD) at intervals of 1-3 months during routine Lung Transplant Clinic follow-up appointments.

Exclusion Criteria:

* UCLA unilateral or bilateral lung transplant recipients, ages: over 65 years of age.
* Females of child bearing age who could become pregnant, refuse to implement appropriate contraception per FDA requirement for "ERA medical treatment" with mandatory MONTHLY monitoring of urine or serum pregnancy tests or become pregnant.
* Concurrent clinically significant chronic liver disease
* Intubated patients
* Patients who cannot perform respiratory maneuvers for office Spirometry and DCO and 6MWD (no tracheostomy).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Estimated); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Measure of FEV1 | Six Months on Therapy
  linearized slopes of loss of lung function (FEV1) / month

SECONDARY OUTCOMES:
Measure of FEV1 | One, Three, Six and Twelve Months
  Absolute change in FEV1
Measure of Six Minute Walk | One, Three, Six and Twelve Months
  Patients' exercise tolerance on six minute walk (6MW) distance
Measure of Pulse Oximetry | One, Three, Six and Twelve Months
  Minimal pulse oximetry saturation (SpO2) during ambulation
Measure of Diffusing Capacity | One, Three, Six and Twelve Months
  Corrected diffusing capacity (DCO)

OTHER OUTCOMES:
BNP Lab Values | One, Three, Six and Twelve Months
  BNP Values
Creatinine Clearance Lab Values | One, Three, Six and Twelve Months
  Creatinine Clearance
Serum Endothelin-1 Lab Values | One, Three, Six and Twelve Months
  Serum Endothelin-1 Values

CONTACTS AND LOCATIONS:
Overall Officials: David J Ross, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of Califonia, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided